CLINICAL TRIAL: NCT03273595
Title: A Prospective, Open-label，Multicentre，Real-word Study of Lapatinib Plus Chemotherapy Versus Trastuzumab Plus Chemotherapy as Neoadjuvant Therapy for Women With HER2-positive and p95HER2-positive，PI3K Mutation，or PTEN Loss Breast Cancer
Brief Title: Lapatinib Plus Chemotherapy Versus Trastuzumab Plus Chemotherapy in HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20162048-1
Record Dates: First submitted 2017-02-22; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2016-06

CONDITIONS: Neoplasms, Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab; Paclitaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Biological: Trastuzumab; Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide
- Experimental group (Experimental)
  Interventions: Drug: Lapatinib; Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Lapatinib
  Arms: Experimental group
Biological: Trastuzumab
  Arms: Control
Drug: Paclitaxel
Drug: Epirubicin
Drug: Cyclophosphamide

SUMMARY:
This is a prospective, open-label, real-word study evaluating the efficacy and safety of lapatinib in combination with chemotherapy versus trastuzumab in combination with chemotherapy in women with HER2-positive and p95HER2-positive ,or PI3K mutation, or PTEN loss breast cancer . Eligible subjects will have newly diagnosed breast cancer (Stage II-III) ; not have received systemic or local treatment . The primary endpoint was the rate of pathological complete response (pCR). The secondary objectives are to evaluate overall survival, overall response rate, clinical benefit response rate and the safety as well as tolerability of lapatinib plus chemotherapy and trastuzumab plus chemotherapy.

Patients will receive lapatinib 1000 mg daily or trastuzumab 4 mg/kg intravenous (IV) load followed by 2 mg/kg IV weekly for a total of 12 weeks. After surgery, patients planned total duration of the anti-HER2 therapy will be one year.

ELIGIBILITY:
Inclusion Criteria:

* Female gender;
* Age ≥18 years;
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
* Histologically confirmed invasive breast cancer:
* Primary tumour greater than 2 cm diameter, measured by clinical examination and mammography or echography,
* p95HER2 positive,or PI3K mutation,or PTEN loss
* Over expression and/or amplification of HER2 in the invasive component of the primary tumour [Wolff et al 2006] and confirmed by a certified laboratory prior to randomisation
* Known hormone receptor status.
* Haematopoietic status:
* Cardiovascular:
* Baseline left ventricular ejection fraction (LVEF) ³ 50% measured by echocardiography (ECHO) or Multiple Gate Acquisition (MUGA) scan,
* Negative serum pregnancy test, within 2-weeks (preferably 7 days) prior to randomization (For women of childbearing potential)
* Fertile patients must use effective contraception (barrier method - condoms, diaphragm - also in conjunction with spermicidal jelly, or total abstinence. Oral, injectable, or implant hormonal contraceptives are not allowed)
* Signed informed consent form (ICF)
* Patient accepts to make available tumour samples for submission to central laboratory to conduct translational studies as part of this protocol

Exclusion Criteria:

* Received any prior treatment for primary invasive breast cancer;
* Previous (less than 10 years) or current history of malignant neoplasms, except for curatively treated:
* Basal and squamous cell carcinoma of the skin;
* Carcinoma in situ of the cervix.
* Patients with a prior malignancy diagnosed more than 10 years prior to randomisation may enter the study. Patients must have been curatively treated with surgery alone. Radiation therapy or systemic therapy (chemotherapy or endocrine) are NOT permitted. Prior diagnoses of breast cancer or melanoma are excluded.
* Diagnosis of inflammatory breast cancer;
* Bilateral cancer;
* This criterion has been deleted from the protocol Version 1. Patients with multi-focal cancer are no longer excluded.
* Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension (≥180/110), unstable diabetes mellitus, dyspnoea at rest, or chronic therapy with oxygen;
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety;
* Unresolved or unstable, serious adverse events from prior administration of another investigational drug;
* Active or uncontrolled infection;
* Dementia, altered mental status, or any psychiatric condition that would prevent the understanding or rendering of ICF;
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded;
* Concurrent neoadjuvant cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy other than the trial therapies);
* Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial;
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trastuzumab or lapatinib or their excipients;
* Pregnant or lactating women;
* Concomitant use of CYP3A4 inhibitors or inducers

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | at the end of week 12

CONTACTS AND LOCATIONS:
Overall Officials: Rui Ling, Doctor, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes